CLINICAL TRIAL: NCT05106127
Title: A Phase 2, Open-Label, Safety Lead-In With Long Term Safety Study of EG-007, Added to the Combination of Lenvatinib Plus Pembrolizumab
Brief Title: Safety Lead-In Study of a Repurposed Drug Added to the Combination of Len Plus Pem
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Evergreen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HPC-EG-007-2.1
Record Dates: First submitted 2021-09-22; First posted 2021-11-03 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Advanced Endometrial Cancer
MeSH Terms: interventions — pembrolizumab; Injections; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EG-007 1000mg + Len + Pem (Experimental): 3 to 6 patients will receive EG-007 1000 mg once weekly starting on the day of injection of Pembrolizimab starting the next 21-day cycle of treatment.
  Interventions: Drug: EG-007; Drug: Pembrolizumab 100 mg/4 mL (25 mg/ml) Injection; Drug: Lenvatinib Capsules
- EG-007 1000mg Loading + Len + Pem (Experimental): 6 to 10 patients will receive EG-007 loading dose of 5000 mg given as 1000 mg daily over 5 consecutive days starting 4 days before the first dose of Pembrolizumab under this protocol.
  Interventions: Drug: EG-007; Drug: Pembrolizumab 100 mg/4 mL (25 mg/ml) Injection; Drug: Lenvatinib Capsules
- EG-007 1000mg D-4 Loading + Len + Pem (Experimental): 6 to 12 patients initiating new regimens of Len+Pem will receive EG-007 loading dose of 5000 mg given as 1000 mg daily over 5 consecutive days starting 4 days before the first dose of Pembrolizumab.
  Interventions: Drug: EG-007; Drug: Pembrolizumab 100 mg/4 mL (25 mg/ml) Injection; Drug: Lenvatinib Capsules

INTERVENTIONS:
Drug: EG-007 — A Repurposed Drug
Drug: Pembrolizumab 100 mg/4 mL (25 mg/ml) Injection — Pembrolizumab will be provided as a sterile, preservative-free, clear to slightly opalescent, colorless to slightly yellow solution that requires dilution for intravenous infusion. Each vial contains 100 mg of pembrolizumab in 4 mL of solution.
Drug: Lenvatinib Capsules — Lenvatinib will be provided as 4-mg and 10-mg capsules. Lenvatinib is formulated with calcium carbonate, mannitol, microcrystalline cellulose, hydroxypropyl cellulose, low-substituted hydroxypropylcellulose, and talc.

SUMMARY:
This is a Phase 2 trial Safety Lead-in trial conducted in 3 cohorts of patients.

A safety lead-in study of the impact of adding the Repurposed Drugs a third agent will be conducted prior to opening enrollment into the compassionate use study. All patients enrolled in the safety lead-in study may continue long-term treatment under this protocol without interruption of dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Female, 18 years and older at the time of informed consent, who has a histologically confirmed diagnosis of endometrial carcinoma, endometroid histology, that is not MSI-H or dMMR ).
2. Documented evidence of advanced (Stage III or IV), or recurrent EC.
3. Must have a recurrence or progressed on a platinum containing chemotherapy regimen and are not candidates for curative surgery or radiation
4. Has historical or fresh tumor biopsy specimen for confirmation of mismatch repair (MMR) status as not MSI-H or dMMR.
5. Has measurable or evaluable disease according to Response Evaluation Criteria In Solid Tumors (RECIST v1.1).
6. Is a candidate for initiation of treatment with the combined regimen of Keytruda plus Lenvima (Len+Pem) OR IS CURRENTLY RECEIVING a tolerated regimen of Len+Pem at the doses specified as the Len+Pem Regimen (per Labeling July 2021)
7. Life expectancy of 12 weeks or more.
8. Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 within 7 days of starting study treatment.
9. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP less than or equal to 150/90 mmHg at screening and no change in antihypertensive medications within 1 week prior to the Cycle 1 Day 1.
10. Adequate renal function defined as creatinine less than or equal to 1.5 × ULN (upper limit of normal) or calculated creatinine clearance greater than or equal to 40 mL/min per the Cockcroft and Gault formula with creatinine levels greater than 1.5 × ULN.

Additional detail upon request.

Exclusion Criteria:

1. Brain metastasis: Previously treated CNS disease needs to be asymptomatic and does not require steroids. Brain metastases must be asymptomatic, fully treated and stable and not requiring steroids within 4 weeks prior to study treatment initiation.
2. Has carcinosarcoma (malignant mixed mullerian tumor), serous carcinoma, endometrial leiomyosarcoma and endometrial stromal sarcomas.
3. Has failed treatment of lenvatinib + pembrolizumab in prior lines of therapy.
4. Except for the allowance of ongoing use of Len+Pem, the protocol excludes patients having received any other prior anticancer treatment within 28 days (or 5 times the half-life time, whichever is shorter) or any investigational agent within 30 days prior to the first dose of study drugs. All acute toxicities related to prior treatments must be resolved to Grade less than or equal to 1.
5. Participants must have recovered adequately from any toxicity and/or complications from major surgery prior to starting therapy.
6. Participants having greater than 1+ proteinuria on urinalysis will undergo 24-h urine collection for quantitative assessment of proteinuria. Participants with urine protein greater than or equal to 1 g/24-hour will be ineligible.
7. Gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of the study drugs
8. Has a pre-existing greater than or equal (>=) Grade 3 gastrointestinal or non-gastrointestinal fistula.
9. Has radiographic evidence of major blood vessel invasion/infiltration.
10. Has clinically significant tumor bleeding within 2 weeks prior to the first dose of study treatment.

Additional detail upon request.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Adverse Events Assessment using CTCAE v5.0 | 1 Cycle of 21 days
  Number of Participants With Treatment-Related Adverse Events as Assessed by NCI CTCAE v5.0, toxicities will be characterized in terms including seriousness, causality, toxicity grading, and action taken with regard to trial treatment. Data Monitoring committee review for safety to proceed through dose escalation.
Tolerability Score measurement using NCI-PRO CTCAE | 1 Cycle of 21 days
  Using NCI-PRO CTCAE to record the tolerability score for patients to evaluate symptomatic toxicities.

SECONDARY OUTCOMES:
Long-term Safety Monitoring for EG-007 plus Len+Pem | At the end of every Cycle (21 days per Cycle), up to 12 Cycles; and upon study exit
  To conduct long-term monitoring of the safety and clinical outcomes for EG-007 plus Len+Pem. The proportion of Participants With Treatment-Related Adverse Events during long-term monitoring.